CLINICAL TRIAL: NCT06570668
Title: Phase 1 Safety, Tolerability and Pharmacokinetics Study of CDD-2101 in Health Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of CDD-2101 in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Chinese Herbal Medicine Drug Development Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDD-2101-P1-6
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: A total of 20 subjects aged 18-65 years with a Body Mass Index (BMI) of 18.5-29.9 kg/m2 will be hospitalized and randomized in a 1:1:1:1:1 ratio (N=4/group) to receive one dose of CDD-2101 at 5, 10, 15 or 20 g and/or placebo by taking a suspension in water orally.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both CDD-2101 and placebo are packed in single-use plain laminated aluminum foil pouches (5 g/sachet). All subjects will take 20 g of granules, i.e. 4 sachets of CDD-2101 and/or placebo, at one time. This will be a double-blind study; group assignment will be blinded to subjects, investigators and all staff involved in the conduct of the study except the unblinded pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 5 g of CDD-2101 and 15 g of placebo; (Experimental): CDD-2101 is a botanical drug candidate in granule form, with same formulation as the Chinese herbal medicine MZRW, based on the water extract from six botanical raw materials (in the form of decoction pieces) including Huomarean, Dahuang, Kuxingren, Houpo, Baishao and Zhishi (stir-fried with wheat bran). Dextrin and magnesium stearate are added as excipients.
  The placebo is in the form of granules for oral use. The granules are a mixture of color and flavor additives (caramel coloring, riboflavin, citric acid and sucrose octaacetate) with dextrin as an excipient.
  Interventions: Drug: CDD-2101
- 10 g of CDD-2101 and 10 g of placebo; (Experimental): CDD-2101 is a botanical drug candidate in granule form, with same formulation as the Chinese herbal medicine MZRW, based on the water extract from six botanical raw materials (in the form of decoction pieces) including Huomarean, Dahuang, Kuxingren, Houpo, Baishao and Zhishi (stir-fried with wheat bran). Dextrin and magnesium stearate are added as excipients.
  The placebo is in the form of granules for oral use. The granules are a mixture of color and flavor additives (caramel coloring, riboflavin, citric acid and sucrose octaacetate) with dextrin as an excipient.
  Interventions: Drug: CDD-2101
- 15 g of CDD-2101 and 5 g of placebo; (Experimental): CDD-2101 is a botanical drug candidate in granule form, with same formulation as the Chinese herbal medicine MZRW, based on the water extract from six botanical raw materials (in the form of decoction pieces) including Huomarean, Dahuang, Kuxingren, Houpo, Baishao and Zhishi (stir-fried with wheat bran). Dextrin and magnesium stearate are added as excipients.
  The placebo is in the form of granules for oral use. The granules are a mixture of color and flavor additives (caramel coloring, riboflavin, citric acid and sucrose octaacetate) with dextrin as an excipient.
  Interventions: Drug: CDD-2101
- 20 g of CDD-2101 (Experimental): CDD-2101 is a botanical drug candidate in granule form, with same formulation as the Chinese herbal medicine MZRW, based on the water extract from six botanical raw materials (in the form of decoction pieces) including Huomarean, Dahuang, Kuxingren, Houpo, Baishao and Zhishi (stir-fried with wheat bran). Dextrin and magnesium stearate are added as excipients.
  Interventions: Drug: CDD-2101
- 20 g of placebo (Placebo Comparator): The placebo is in the form of granules for oral use. The granules are a mixture of color and flavor additives (caramel coloring, riboflavin, citric acid and sucrose octaacetate) with dextrin as an excipient.
  Interventions: Drug: CDD-2101

INTERVENTIONS:
Drug: CDD-2101 — All subjects will receive 4 sachets of CDD-2101 and/or placebo at a time based on the computer-generated randomization. An unblinded pharmacist will mix the assigned dose of CDD-2101 and/or placebo with 400 mL of water at 70-80°C, cool it to a comfortable temperature and keep it at room temperature for not longer than 1 h. A blinded study nurse or investigator will dispense the suspension to the assigned subject. The subject will drink it under supervision within 15 minutes.

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single-dose study to confirm the safety, tolerability and pharmacokinetic profile of CDD-2101 in healthy subjects. A total of 20 subjects aged 18-65 years with a Body Mass Index (BMI) of 18.5-29.9 kg/m2 will be hospitalized and randomized in a 1:1:1:1:1 ratio (N=4/group) to receive one dose of CDD-2101 at 5, 10, 15 or 20 g and/or placebo by taking a suspension in water orally. Subjects will complete a daily bowel habit diary 7 days and refrain from food containing any of the botanicals in CDD-2101 for at least 3 days prior to randomization. Subjects will also need to abstain from the consumption of any xanthine containing products (e.g. coffee, tea, chocolate, or Coca-Cola like drinks) more than 6 cups per day (or equivalent) 24 hours before randomization. A 12-lead electrocardiogram (ECG) and a full physical examination will be performed at pre-dose and 24 h post-dose. Blood samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 h post-dose. Urine samples will be collected immediately before and at 0-3 h, 3-6 h, 6-9 h, 9-12 h and 12-24 h post-dose. Vital signs will be measured at 0 (pre-dose), 1, 2, 3, 4, 8, 12 and 24 h post-dose. Adverse events (AEs) will be monitored during the study period. After the 24 h post-dose procedures are completed, the investigator will confirm the subjects are in good health before discharging them. All subjects will have a follow-up visit 3 days after the dose of investigational drug. Plasma samples will be analyzed for complete blood count, liver and kidney function markers, total cholesterol, glucose, calcium and marker compounds of CDD-2101. Urine samples will be processed for quantitation of marker compounds of CDD-2101. The primary endpoint will be safety and tolerability of CDD-2101, with vital signs, reported number and seriousness of AEs, physical examination, and laboratory tests as outcome measures. The secondary endpoints will be the pharmacokinetic profile, with outcome measures including peak plasma concentration (Cmax), time to reach Cmax (Tmax), area under the curve (AUC) from 0 to 24 h post-dose and renal excretion of marker compounds, and bowel movement with the number of complete spontaneous bowel movement (CSBM) and stool quality based on the Bristol Stool Form Scale as outcome measures.

DETAILED DESCRIPTION:
A total of 20 eligible healthy subjects aged 18-65 years, body weight of 50kg or more with a BMI of 18.5-29.9 kg/m2 will be hospitalized and randomized in a 1:1:1:1:1 ratio (N=4/group) to receive one dose of CDD-2101 at 5, 10, 15 or 20 g and/or placebo by taking a suspension in water orally.

All subjects will be required to refrain from food containing any of the botanicals in CDD-2101 for at least 3 days prior to randomization.

Each subject will also be required to complete a daily bowel habit diary logging all clinical events during the study. The diary may be completed online using an electronic case report form (eCRF) or by pen and paper. Each subject will be provided with the study diary after the screening visit. Subjects will be instructed to record in the diary every day, including the day admitted to the CPU, and continue until 3 days after the dose of investigational drug.

Study diary will be collected and reviewed for completeness at baseline/randomization, and at the end-of-follow-up visit (Day 3). Authorized study personnel will transcribe all data collected from the physical diaries into eCRF. All information collected from the diaries will be analyzed for primary and secondary endpoints in the study.

All subjects will be instructed about diary completion at every study visit. Documentation that subjects have been appropriately instructed (and re-instructed as necessary) on diary completion should be recorded in the subject's source notes.

Subjects who are not consistent or thorough with study diary completion may receive phone reminders if deemed necessary by the investigators. The authorized study personnel providing phone reminders must document the phone contact process in the subject's source notes.

A sample of the diary is in Appendix 1. The diary is to record the number of bowel openings, a sense of complete/incomplete evacuation, and quality of stool according to the Bristol Stool Form Scale (Appendix 2). The Bristol Stool Form Scale is a medical aid designed to classify stools into seven groups and will be supplied to the subjects.

Bristol Stool Form Scale is defined as 7-point scale in which a score of 1 - separate hard lumps, 2 - sausage shaped but lumpy, 3 - sausage-like with cracks on the surface, 4 - sausage-like but smooth and soft, 5 - soft blobs with clearcut edge, 6 - fluffy pieces with ragged edges ragged edges, and 7 - watery with no solid pieces.

A 12-lead ECG will be performed at pre-dose and 24 h post-dose. Full physical examination will be performed 24 h post-dose. Blood samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 2, 4, 8, 12 and 24 h post-dose. Urine samples will be collected immediately before and at 0-3, 3-6, 6-9, 9-12 and 12-24 h post-dose. Vital signs will be assessed at 0 (pre-dose), 1, 2, 3, 4, 8, 12 and 24 h post-dose. AEs will be monitored during the study period. Upon completion of the 24 h post-dose procedures, the investigator will confirm that it is safe (i.e., the subject appears healthy) before discharging the participants. All subjects will return for a follow-up visit on Day 4 after the last dose of investigational drug.

The primary endpoint will be safety and tolerability of CDD-2101, with vital signs, reported number and seriousness of AEs, physical examination, and laboratory tests as outcome measures.

The secondary endpoint will be the pharmacokinetic profile with Cmax, Tmax, AUC from 0 to 24 h post-dose and renal excretion as outcome measures, and bowel movement with the number of CSBM and stool quality based on the Bristol Stool Form Scale as outcome measures.

Available data will be entered in a secure clinical database using eCRF, along with subject information.

ELIGIBILITY:
Inclusion Criteria:

* An individual must meet all the criteria below to be eligible for participation in this study:

  1. Male or female
  2. Aged 18-65 years (inclusive)
  3. Body weight of 50kg or more
  4. BMI 18.5-29.9 kg/m2 (inclusive)
  5. Normal hepatic: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and gamma glutamyl transferase (GGT) and total bilirubin not elevated more than 1.2-fold above the upper limit of normal (ULN)
  6. Normal renal function: glomerular filtration rate (GFR) ≥ 90 mL/min/1.7m2
  7. Understand the study procedures and agree to participate by providing written informed consent
  8. Be willing and able to comply with all study procedures and restrictions
  9. Be a nonsmoker who has not used tobacco- or nicotine-containing products (e.g., nicotine patch) for at least 6 months before administration of the investigational drug
  10. Be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead ECG, and vital sign assessment performed at the Screening Visit and before administration of the investigational drug
  11. Contraceptive use by men or women should be consistent with local regulations regarding the methods of conception for those participating in clinical study

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded:

  1. Pregnant, trying to become pregnant or lactating
  2. Use of any prescription, non-prescription drug and investigational drug within 30 days prior to administration of the study drug
  3. Has a substance abuse disorder
  4. Has a history of clinically significant endocrine, gastrointestinal (including motility disorder and intestinal obstruction), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
  5. Has a history of cancer (malignancy)
  6. Has a known hypersensitivity to any component of the formulation of CDD-2101, its related compounds or placebo, or allergy to Chinese herbal medicine
  7. Has a history of significant multiple and/or severe allergies (e.g., food, drug or latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food
  8. Had major surgery, donated, or lost 1 unit of blood (approximately 500 mL) within 8 weeks before administration of the investigational drug
  9. Diagnosis of bowel disorders based on the Rome IV criteria
  10. Has a history of positive for hepatitis B, hepatitis C or HIV
  11. Has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink is approximately equivalent to: beer (354 mL/12 ounces), wine (118 mL/4 ounces), or distilled spirits (29.5 mL/1 ounce)
  12. Has participated in another investigational trial within 4 weeks before the pretrial (Screening) visit. The 4-week window will be derived from the date of the last trial procedure and/or AE related to the trial procedure in the previous trial to the pretrial/Screening Visit of the current trial.
  13. Is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the sponsor or Contract Research Organization (CRO)
  14. Having received another investigational drug or been participated in an investigational drug or device study within 30 days before administration of the investigational drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
potential AEs | baseline, pre-intervention, randomization, follow-up 4 days after randomization, through study completion, i.e. from screening till complete follow up visit which is about 26 days
  based on the changes of vital signs, 12-leads ECG, clinical laboratory results and physical examinations

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] - cannabisin B | pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum plasma concentration [Cmax] - rhein | pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum plasma concentration [Cmax] - magnolol | pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum plasma concentration [Cmax] - paeoniflorin | pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum plasma concentration [Cmax] - albiflorin | pre-dose, and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum plasma concentration [Cmax] - synephrine | pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - cannabisin B | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - rhein | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - aloe emodin | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - amygdalin | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - magnolol | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - honokiol | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - paeoniflorin | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - albiflorin | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.
Maximum urine concentration [Cmax] - synephrine | pre-dose and at 0-3, 3-6, 6-9, 9-12 and 12-24 hours after dose
  The marker compounds will be calculated by establishing curves of each analyte.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial Inc, Newark, New Jersey, United States